CLINICAL TRIAL: NCT03867110
Title: A Phase 3, Double-Blind Efficacy and Safety Study of Ezetimibe (SCH 58235) 10 mg in Addition to Atorvastatin Compared to Placebo in Subjects With Primary Hypercholesterolemia (Protocol P00692)
Brief Title: An Efficacy and Safety Study of Ezetimibe (MK-0653, SCH 58235) in Addition to Atorvastatin Compared to Placebo in Participants With Primary Hypercholesterolemia (MK-0653-013)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P00692; MK-0653-013 (Other: Merck Protocol Number); P00692 (Other: Schering-Plough Protocol Number)
Record Dates: First submitted 2019-03-06; First posted 2019-03-07 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
Keywords: Hypercholesterolemia; Ezetimibe; Atorvastatin; Low density lipoprotein-cholesterol
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Placebo (Placebo Comparator): Placebo is to be taken orally once a day (QD) in the morning for 12 consecutive weeks.
  Interventions: Drug: Placebo
- Ezetimibe 10 mg (Active Comparator): Ezetimibe 10 mg (MK-0653, SCH 58235) is to be taken orally QD in the morning for 12 consecutive weeks.
  Interventions: Drug: Ezetimibe 10 mg
- Atorvastatin 10 mg (Active Comparator): Atorvastatin 10 mg is to be taken orally QD in the morning for 12 consecutive weeks.
  Interventions: Drug: Atorvastatin 10 mg
- Ezetimibe 10 mg + Atorvastatin 10 mg (Experimental): Ezetimibe 10 mg (MK-0653, SCH 58235) + Atorvastatin 10 mg is to be taken orally QD in the morning for 12 consecutive weeks.
  Interventions: Drug: Ezetimibe 10 mg; Drug: Atorvastatin 10 mg
- Atorvastatin 20 mg (Active Comparator): Atorvastatin 20 mg is to be taken orally QD in the morning for 12 consecutive weeks.
  Interventions: Drug: Atorvastatin 20 mg
- Ezetimibe 10 mg + Atorvastatin 20 mg (Experimental): Ezetimibe 10 mg (MK-0653, SCH 58235) + Atorvastatin 20 mg is to be taken orally QD in the morning for 12 consecutive weeks.
  Interventions: Drug: Ezetimibe 10 mg; Drug: Atorvastatin 20 mg
- Atorvastatin 40 mg (Active Comparator): Atorvastatin 40 mg is to be taken orally QD in the morning for 12 consecutive weeks.
  Interventions: Drug: Atorvastatin 40 mg
- Ezetimibe 10 mg + Atorvastatin 40 mg (Experimental): Ezetimibe 10 mg (MK-0653, SCH 58235) + Atorvastatin 40 mg is to be taken orally QD in the morning for 12 consecutive weeks.
  Interventions: Drug: Ezetimibe 10 mg; Drug: Atorvastatin 40 mg
- Atorvastatin 80 mg (Active Comparator): Atorvastatin 80 mg is to be taken orally QD in the morning for 12 consecutive weeks.
  Interventions: Drug: Atorvastatin 80 mg
- Ezetimibe 10 mg + Atorvastatin 80 mg (Experimental): Ezetimibe 10 mg (MK-0653, SCH 58235) + Atorvastatin 80 mg is to be taken orally QD in the morning for 12 consecutive weeks.
  Interventions: Drug: Ezetimibe 10 mg; Drug: Atorvastatin 80 mg

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: Ezetimibe 10 mg
  Other Names: MK-0653; SCH 58235; ZETIA®
  Arms: Ezetimibe 10 mg; Ezetimibe 10 mg + Atorvastatin 10 mg; Ezetimibe 10 mg + Atorvastatin 20 mg; Ezetimibe 10 mg + Atorvastatin 40 mg; Ezetimibe 10 mg + Atorvastatin 80 mg
Drug: Atorvastatin 10 mg
  Other Names: LIPITOR®
  Arms: Atorvastatin 10 mg; Ezetimibe 10 mg + Atorvastatin 10 mg
Drug: Atorvastatin 20 mg
  Other Names: LIPITOR®
  Arms: Atorvastatin 20 mg; Ezetimibe 10 mg + Atorvastatin 20 mg
Drug: Atorvastatin 40 mg
  Other Names: LIPITOR®
  Arms: Atorvastatin 40 mg; Ezetimibe 10 mg + Atorvastatin 40 mg
Drug: Atorvastatin 80 mg
  Other Names: LIPITOR®
  Arms: Atorvastatin 80 mg; Ezetimibe 10 mg + Atorvastatin 80 mg

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, balanced-parallel-group, efficacy and safety trial of ezetimibe coadministered with atorvastatin in adult participants with primary hypercholesterolemia. The primary hypothesis is that the coadministration of ezetimibe 10 mg/day with atorvastatin (pooled across all doses: 10 mg, 20 mg, 40 mg, 80 mg) will result in a significantly greater reduction in direct low density lipoprotein-cholesterol (LDL-C) when compared with atorvastatin (pooled across all doses: 10 mg, 20 mg, 40 mg, 80 mg) alone and ezetimibe 10 mg alone.

ELIGIBILITY:
Inclusion Criteria:

* If female, is not pregnant or breastfeeding, and is either not a woman of childbearing potential (WOCBP), or is a WOCBP who has used a contraceptive consistent with local regulations.
* Postmenopausal women who are receiving postmenopausal hormonal therapy or raloxifene must be maintained on a stable estrogen (ERT), estrogen/progestin (HRT) or raloxifene regimen during the study period.
* Primary hypercholesterolemic participants with a plasma LDL-Cholesterol ≥145 mg/dL (3.75 mmol/L) and ≤250 mg/dL (6.48 mmol/L) and plasma triglyceride ≤350 mg/dL (3.99 mmol/L) after adequate drug washout
* Must be willing to observe the National Cholesterol Education Program (NCEP) Step I diet as determined by a Ratio of Ingested Saturated fat and Cholesterol to Calories (RISCC) score not greater than 24 throughout this study. Ability to complete Diet Diaries needs to be demonstrated.

Exclusion Criteria:

* Has a history of mental instability, drug/alcohol abuse within the past 5 years, or major psychiatric illness not adequately controlled and stable on pharmacotherapy.
* Underlying disease likely to limit life span to less than 1 year.
* Participants with hypercholesterolemia in whom withholding of approved lipid-lowering therapy would be inappropriate.
* Have previously been randomized in any of the studies evaluating Ezetimibe (SCH 58235).
* Known hypersensitivity or any contraindication to atorvastatin (LIPITOR®).
* Pregnant or lactating women.
* Congestive heart failure New York Heart Association (NYHA) Class III or IV.
* Uncontrolled cardiac arrhythmias.
* Myocardial infarction, coronary bypass surgery or angioplasty within 6 months of study entry.
* Unstable or severe peripheral artery disease within 3 months of study entry.
* Unstable angina pectoris.
* Disorders of the hematologic, digestive or central nervous systems including cerebrovascular disease and degenerative disease that would limit study evaluation or participation.
* Uncontrolled or newly diagnosed (within 1 month of study entry) diabetes mellitus.
* Uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoproteins.
* Known impairment of renal function (plasma creatinine >2.0 mg/dL), dysproteinemia, nephrotic syndrome or other renal disease.
* Active or chronic hepatobiliary or hepatic disease.
* Participants who are known to be Human Immunodeficiency Virus (HIV) positive.
* Participants with known coagulopathy.
* Lipid-altering agents, other than study drugs for the whole duration of the study.
* Oral corticosteroids.
* Cardiovascular drugs such as: beta blockers, calcium channel blockers, ACE inhibitors, nitrates or α-adrenergic blockers or thiazide diuretics will be allowed, provided the dose remains constant for the duration of the study and the participant has received a stable dose for at least 8 weeks before the initial qualifying LDL-C level is drawn. Aspirin up to 325 mg/day is permitted. In addition, aspirin is allowed as a as needed (prn) concomitant medication.
* Treatment with psyllium or other fiber-based laxatives unless treated with a stable regimen for at least 4 weeks before initial qualifying lipid determination. Dose must remain constant throughout the study period.
* Treatment with troglitazone (Rezulin®) unless treated with a stable regimen for at least 6 weeks before initial qualifying lipid determination. Dose must remain constant throughout the study period.
* Treatment with cyclosporine.
* Use of any investigational drugs within 30 days of study entry.
* Treatment with agents with known drug interaction with atorvastatin including antifungal azoles (itraconazole and ketoconazole), macrolide antibiotics (erythromycin and clarithromycin), and nefazodone. In addition, treatment with other agents that may interfere with or induce the CYP3A4 isoenzyme of the cytochrome P450 system should be avoided.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 628 (Actual)
Dates: Start 2000-03-06 (Actual); Primary Completion 2001-07-27 (Actual); Study Completion 2001-07-27 (Actual)

PRIMARY OUTCOMES:
Percent Change from Baseline at Week 12 of Plasma Low Density Lipoprotein Cholesterol (LDL-C) | Baseline and Week 12
  Plasma LDL-C determined following a standard ultracentrifugation / precipitation (quantification) procedure (direct LDL-C). Participants had LDL-C levels assessed at baseline and after 12 weeks of study drug administration. The percent change from baseline was calculated.

SECONDARY OUTCOMES:
Percent Change from Baseline at Week 12 for Calculated Low Density Lipoprotein-Cholesterol (LDL-C) | Baseline and Week 12
  Participants had LDL-C levels assessed at baseline and after 12 weeks of study drug administration. The percent change from baseline was calculated.
Percent Change from Baseline at Week 12 for Total Cholesterol (TC) | Baseline and Week 12
  Participants had TC levels assessed at baseline and after 12 weeks of study drug administration. The percent change from baseline was calculated.
Percent Change from Baseline at Week 12 for Triglycerides (TG) | Baseline and Week 12
  Participants had TG levels assessed at baseline and after 12 weeks of study drug administration. The percent change from baseline was calculated.
Percent Change from Baseline at Week 12 for High Density-Lipoprotein-Cholesterol (HDL-C) | Baseline and Week 12
  Participants had HDL-C levels assessed at baseline and after 12 weeks of study drug administration. The percent change from baseline was calculated.
Percent Change from Baseline at Week 12 for Apolipoprotein B (Apo B) | Baseline and Week 12
  Participants had Apo B levels assessed at baseline and after 12 weeks of study drug administration. The percent change from baseline was calculated.
Percent Change from Baseline at Week 12 for Non-High Density-Lipoprotein-Cholesterol (Non-HDL-C) | Baseline and Week 12
  Participants had Non-HDL-C levels assessed at baseline and after 12 weeks of study drug administration. The percent change from baseline was calculated.
Percent Change from Baseline at Week 12 for High Density-Lipoprotein 2-Cholesterol (HDL2-C) | Baseline and Week 12
  Participants had HDL2-C levels assessed at baseline and after 12 weeks of study drug administration. The percent change from baseline was calculated.
Percent Change from Baseline at Week 12 for High Density-Lipoprotein 3-Cholesterol (HDL3-C) | Baseline and Week 12
  Participants had HDL3-C levels assessed at baseline and after 12 weeks of study drug administration. The percent change from baseline was calculated.
Percent Change from Baseline at Week 12 for Apolipoprotein A-I (Apo A-I), | Baseline and Week 12
  Participants had Apo A1 levels assessed at baseline and after 12 weeks of study drug administration. The percent change from baseline was calculated.
Percent Change from Baseline at Week 12 for Direct Low Density-Lipoprotein 3-Cholesterol/High Density-Lipoprotein 3-Cholesterol (LDL-C/HDL-C) Ratio | Baseline and Week 12
  Participants had LDL-C and HDL-C levels assessed at baseline and after 12 weeks of study drug administration. The percent change from baseline in the LDL-C/HDL-C ratio was calculated.
Percent Change from Baseline at Week 12 for Direct Total Cholesterol/High Density-Lipoprotein 3-Cholesterol (TC/HDL-C) Ratio | Baseline and Week 12
  Participants had TC and HDL-C levels assessed at baseline and after 12 weeks of study drug administration. The percent change from baseline in the TC/HDL-C ratio was calculated.
Percent Change from Baseline at Week 12 for Lipoprotein (a) (Lp[a]) | Baseline and Week 12
  Participants had Lp(a) levels assessed at baseline and after 12 weeks of study drug administration. The percent change from baseline was calculated.
The Percentage of Participants Achieving National Cholesterol Education Program (NCEP) Adult Treatment Panel (ATP II) Target Goal for Direct Low Density Lipoprotein-Cholesterol (LDL-C) | Week 12
  LDL cholesterol level goal is <100 mg per deciliter (2.60 mmol per L)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ballantyne CM, Houri J, Notarbartolo A, Melani L, Lipka LJ, Suresh R, Sun S, LeBeaut AP, Sager PT, Veltri EP; Ezetimibe Study Group. Effect of ezetimibe coadministered with atorvastatin in 628 patients with primary hypercholesterolemia: a prospective, randomized, double-blind trial. Circulation. 2003 May 20;107(19):2409-15. doi: 10.1161/01.CIR.0000068312.21969.C8. Epub 2003 Apr 28. PMID 12719279